CLINICAL TRIAL: NCT07238699
Title: An Evaluation of the Safety and Tolerability of Ocular Lubricants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DEE253-E003
Record Dates: First submitted 2025-11-17; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease
Keywords: Itchy eyes; Stinging eyes; Scratchy eyes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: FID123440, then FID123437 (Experimental): One drop of FID123440 test formulation in each eye in Period 1, followed by 1 drop of FID123437 test formulation in each eye in Period 2 as randomized. Each period is 1 day long with at least 2 calendar days separating the periods.
  Interventions: Other: FID123440 test formulation; Other: FID123437 test formulation
- Sequence 2: FID123437, then FID123440 (Experimental): One drop of FID123437 test formulation in each eye in Period 1, followed by 1 drop of FID123440 test formulation in each eye in Period 2 as randomized. Each period is 1 day long with at least 2 calendar days separating the periods.
  Interventions: Other: FID123437 test formulation; Other: FID123440 test formulation

INTERVENTIONS:
Other: FID123440 test formulation — Investigational product
  Arms: Sequence 1: FID123440, then FID123437
Other: FID123437 test formulation — Investigational product
Other: FID123440 test formulation — Investigational product
  Arms: Sequence 2: FID123437, then FID123440

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of two new artificial tear formulations in subjects with moderate dry eye disease.

DETAILED DESCRIPTION:
Each subject will receive 2 investigational products (one drop per eye of each investigational product) in a cross-over study design according to a randomization schedule. Individual duration of participation will be approximately 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing and able to understand and sign an ethics committee approved informed consent form.
* Subject must be willing and able to attend all study visits as required by the protocol.
* Subject must exhibit symptoms of dry eye at the Screening Visit.
* Subject must currently use artificial tears.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has any known active ocular disease and/or infection.
* Has any known infection or inflammation that requires treatment or has a systemic condition that, in the opinion of the investigator, may affect a study outcome variable.
* Any ocular injury to either eye in the 12 weeks prior to screening.
* Current wearer of contact lenses or has a history of contact lens wear within the previous 1 month.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) | Visit 2 [1 to 7 days after Visit 1/Screening (Day 1)] through Exit Visit. Exit Visit will occur 3 to 13 days after Visit 2 depending on observed visit windows.]
  An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). The number of adverse events as observed or reported will be recorded.
Number of Subjects with Biomicroscopy Findings Outside of Normal Limit | Visit 1/Screening (Day 1) through Exit Visit. Exit Visit will occur 4 to 20 days after Visit 1 depending on observed visit windows.
  The investigator will observe the corneal and other ocular structures under white light of the slit lamp. The number of subjects with biomicroscopy findings outside of normal limits will be recorded.
Best Corrected Visual Acuity (BCVA) | Visit 1/Screening (Day 1) through Exit Visit. Exit Visit will occur 4 to 20 days after Visit 1 depending on observed visit windows.
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) letter charts and recorded in logarithm Minimum angle of resolution (logMar).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (5):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States
- Australia (4):
  - School of Optometry and Vision, Sydney, New South Wales
  - Ophthalmic Trials Australia, Teneriffe, Queensland
  - The University of Melbourne, Department of Optometry and Vision Science, Carlton, Victoria
  - Deakin Collaborative Eye Care Clinic, Deakin University, Waurn Ponds, Victoria